CLINICAL TRIAL: NCT01343888
Title: A Phase III, Randomised, Double-blind and Placebo-controlled Study of Once Daily BI 201335 120 mg for 12 or 24 Weeks or BI 201335 240 mg for 12 Weeks in Combination With Pegylated Interferon-alpha and Ribavirin in Treatment-naïve Patients With Genotype 1 Chronic Hepatitis C Infection
Brief Title: Efficacy and Safety of BI 201335 (Faldaprevir) in Combination With Pegylated Interferon-alpha and Ribavirin in Treatment-naïve Genotype 1 Hepatitis C Infected Patients (STARTverso 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.30; 2010-021716-42 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-20; First posted 2011-04-28 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — faldaprevir

ARMS (3):
- PegIFN/RBV (Active Comparator): PegIFN/RBV for 48 weeks
  Interventions: Drug: PegIFN/RBV
- BI 201335 for 12 or 24 weeks (Experimental): BI 201335 once daily low dose for 12 or 24 weeks in combination with PegIFN/RBV for 24 or 48 weeks
  Interventions: Drug: PegIFN/RBV; Drug: BI 201335
- Placebo and PegIFN/RBV (Active Comparator): Placebo (oral) once daily plus PegIFN/RBV (subcutaneous injection/oral) for 24 weeks, followed by PegIFN/RBV alone up to Week 48.
  Interventions: Drug: PegIFN/RBV; Drug: Placebo

INTERVENTIONS:
Drug: PegIFN/RBV — PegIFN/RBV for 48 weeks
Drug: BI 201335 — BI 201335 once daily high dose
  Arms: BI 201335 for 12 or 24 weeks
Drug: BI 201335 — BI 201335 once daily low dose
  Arms: BI 201335 for 12 or 24 weeks
Drug: Placebo
  Arms: Placebo and PegIFN/RBV

SUMMARY:
The objective of this trial is to evaluate the efficacy and safety of two different treatment regimens with BI 201335, both in combination with PegIFN/RBV) as compared to standard of care (SOC) with PegIFN/RBV alone.

ELIGIBILITY:
Inclusion criteria:

1. Chronic hepatitis C infection, diagnosed by positive anti-HCV antibodies and detected HCV RNA at screening in addition to:

   1. positive anti-HCV antibodies or detected HCV RNA at least 6 months prior to screening; or,
   2. liver biopsy consistent with chronic HCV infection.
2. HCV genotype 1 infection confirmed by genotypic testing at screening.
3. Therapy-naïve to interferon, pegylated interferon, ribavirin or any antiviral / immunomodulatory drug for acute or chronic HCV infection.
4. HCV RNA = 1,000 IU/mL at screening
5. Documentation of a liver biopsy within 3 years or fibroscan within 6 months prior to randomization.

   Note: If cirrhosis has been previously demonstrated on a biopsy, then biopsies obtained more than 3 years before randomization need not be repeated. Biopsies may be waived for patients who would be placed at risk from the procedure. Inability to do a liver biopsy in patients at risk for the procedure should not exclude such patients from a trial.
6. Age 18 to 70 years
7. Female patients:

   1. with documented hysterectomy,
   2. who have had both ovaries removed,
   3. with documented tubal ligation,
   4. who are post-menopausal with last menstrual period at least 12 months prior to screening, or
   5. of childbearing potential with a negative serum pregnancy test at screening and Day 1, that, if sexually active, agree to use one of the appropriate medically accepted methods of birth control from the date of screening until 7 months after the last dose of ribavirin in addition to the consistent and correct use of a condom. Patients must agree not to breast-feed at any time from the date of screening until 7 months after the last dose of ribavirin.

   Medically accepted methods of contraception for females in this trial are ethinyl estradiol containing contraceptives, diaphragm with spermicide substance and intra-uterine device.

   Male patients:
   1. who are documented to be sterile, or
   2. who are without pregnant female partner(s) and consistently and correctly use a condom while their female partner(s) (if of child-bearing potential) use one of the appropriate medically accepted methods of birth control from the date of screening until 7 months after the last dose of ribavirin. It is in the responsibility of the male patient to ensure that his partner(s) is not pregnant prior to screening into the study or becomes pregnant during the treatment and the observation phase. Female partners of childbearing potential should perform monthly pregnancy tests from the date of screening until 7 months after the last dose of ribavirin (tests will be provided by the sponsor).
8. Signed informed consent form prior to trial participation

Exclusion criteria:

1. HCV infection of mixed genotype (1/2, 1/3, and 1/4) diagnosed by genotypic testing at screening
2. Evidence of acute or chronic liver disease due to causes other than chronic HCV infection. Incidental steatosis diagnosed by biopsy is not an exclusion criterion.
3. HIV co-infection
4. Hepatitis B virus (HBV) infection based on presence of HBs-Ag
5. Active malignancy, or history of malignancy within the last 5 years prior to screening (with an exception of appropriately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix)
6. Active or, history of alcohol or illicit drug abuse other than cannabis within the past 12 months
7. A condition that is defined as one which in the opinion of investigator may put the patient at risk because of participation in this study, may influence the results of this study, or limit the patients ability to participate in this study
8. Usage of any investigational drugs within 30 days prior to screening, or planned usage of an investigational drug during the course of this study.
9. Received concomitant systemic antiviral, hematopoietic growth factor, or immunomodulatory treatment within 30 days prior to randomization. Patients being treated with oral antivirals such as acyclovir, famciclovir or valacyclovir for recurrent herpes simplex infection; or with oseltamivir or zanamivir for influenza A infection, may be screened.
10. Received silymarin (milk thistle), glycyrrhizin, or Sho-saiko-to (SST) within 28 days prior to randomization and throughout the treatment phase of this trial.
11. Known hypersensitivity to any ingredient of the study drugs.
12. Alpha fetoprotein value > 100 ng/mL at screening; if > 20 ng/mL and = 100 ng/mL, patients may be included if there is no evidence of liver cancer in an appropriate imaging study (e.g., ultrasound, CT scan, or MRI) within last 6 months prior to randomization (Visit 2).

Other exclusion criteria related to pegylated interferon and/or ribavirin restrictions are not listed here.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2011-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (98):
- Austria (4):
  - 1220.30.4303 Boehringer Ingelheim Investigational Site, Linz
  - 1220.30.4301 Boehringer Ingelheim Investigational Site, Vienna
  - 1220.30.4302 Boehringer Ingelheim Investigational Site, Vienna
  - 1220.30.4304 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (6):
  - 1220.30.3201 Boehringer Ingelheim Investigational Site, Brussels
  - 1220.30.3207 Boehringer Ingelheim Investigational Site, Brussels
  - 1220.30.3204 Boehringer Ingelheim Investigational Site, Edegem
  - 1220.30.3205 Boehringer Ingelheim Investigational Site, Ghent
  - 1220.30.3202 Boehringer Ingelheim Investigational Site, Leuven
  - 1220.30.3203 Boehringer Ingelheim Investigational Site, Liège
- France (12):
  - 1220.30.3314 Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 1220.30.3301 Boehringer Ingelheim Investigational Site, Clichy
  - 1220.30.3311 Boehringer Ingelheim Investigational Site, Lille
  - 1220.30.3303 Boehringer Ingelheim Investigational Site, Marseille
  - 1220.30.3304 Boehringer Ingelheim Investigational Site, Montpellier
  - 1220.30.3305 Boehringer Ingelheim Investigational Site, Nice
  - 1220.30.3302 Boehringer Ingelheim Investigational Site, Paris
  - 1220.30.3309 Boehringer Ingelheim Investigational Site, Paris
  - 1220.30.3316 Boehringer Ingelheim Investigational Site, Pessac
  - 1220.30.3315 Boehringer Ingelheim Investigational Site, Rennes
  - 1220.30.3312 Boehringer Ingelheim Investigational Site, Saint-Laurent-du-Var
  - 1220.30.3313 Boehringer Ingelheim Investigational Site, Toulouse
- Germany (16):
  - 1220.30.4917 Boehringer Ingelheim Investigational Site, Aachen
  - 1220.30.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.30.4904 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.30.4916 Boehringer Ingelheim Investigational Site, Bonn
  - 1220.30.4913 Boehringer Ingelheim Investigational Site, Dortmund
  - 1220.30.4906 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1220.30.4909 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1220.30.4912 Boehringer Ingelheim Investigational Site, Erlangen
  - 1220.30.4901 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1220.30.4908 Boehringer Ingelheim Investigational Site, Hamburg
  - 1220.30.4907 Boehringer Ingelheim Investigational Site, Herne
  - 1220.30.4914 Boehringer Ingelheim Investigational Site, Kiel
  - 1220.30.4903 Boehringer Ingelheim Investigational Site, Leipzig
  - 1220.30.4911 Boehringer Ingelheim Investigational Site, Mainz
  - 1220.30.4905 Boehringer Ingelheim Investigational Site, München
  - 1220.30.4915 Boehringer Ingelheim Investigational Site, Ulm
- Japan (20):
  - 1220.30.8106 Boehringer Ingelheim Investigational Site, Chiba, Chiba
  - 1220.30.8111 Boehringer Ingelheim Investigational Site, Gifu, Gifu
  - 1220.30.8107 Boehringer Ingelheim Investigational Site, Itabashi-ku, Tokyo
  - 1220.30.8112 Boehringer Ingelheim Investigational Site, Izunokuni, Shizuoka
  - 1220.30.8108 Boehringer Ingelheim Investigational Site, Kamakura, Kanagawa
  - 1220.30.8117 Boehringer Ingelheim Investigational Site, Kita-gun, Kagawa
  - 1220.30.8109 Boehringer Ingelheim Investigational Site, Kofu, Yamanashi
  - 1220.30.8116 Boehringer Ingelheim Investigational Site, Kurashiki, Okayama
  - 1220.30.8118 Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - 1220.30.8110 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 1220.30.8113 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1220.30.8105 Boehringer Ingelheim Investigational Site, Namegata, Ibaraki
  - 1220.30.8114 Boehringer Ingelheim Investigational Site, Nishinomiya, Hyogo
  - 1220.30.8119 Boehringer Ingelheim Investigational Site, Omura, Nagasaki
  - 1220.30.8122 Boehringer Ingelheim Investigational Site, Omuta, Fukuoka
  - 1220.30.8121 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1220.30.8101 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1220.30.8102 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1220.30.8115 Boehringer Ingelheim Investigational Site, Tanabe, Wakayama
  - 1220.30.8104 Boehringer Ingelheim Investigational Site, Tsuchiura, Ibaraki
- Portugal (8):
  - 1220.30.3503 Boehringer Ingelheim Investigational Site, Aveiro
  - 1220.30.3509 Boehringer Ingelheim Investigational Site, Barreiro
  - 1220.30.3506 Boehringer Ingelheim Investigational Site, Coimbra
  - 1220.30.3501 Boehringer Ingelheim Investigational Site, Lisbon
  - 1220.30.3505 Boehringer Ingelheim Investigational Site, Lisbon
  - 1220.30.3507 Boehringer Ingelheim Investigational Site, Lisbon
  - 1220.30.3502 Boehringer Ingelheim Investigational Site, Porto
  - 1220.30.3504 Boehringer Ingelheim Investigational Site, Vila Real
- Romania (4):
  - 1220.30.4001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1220.30.4002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1220.30.4003 Boehringer Ingelheim Investigational Site, Bucharest
  - 1220.30.4004 Boehringer Ingelheim Investigational Site, Bucharest
- Russia (6):
  - 1220.30.7002 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1220.30.7001 Boehringer Ingelheim Investigational Site, Moscow
  - 1220.30.7004 Boehringer Ingelheim Investigational Site, Moscow
  - 1220.30.7005 Boehringer Ingelheim Investigational Site, Moscow
  - 1220.30.7006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1220.30.7007 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Spain (8):
  - 1220.30.3406 Boehringer Ingelheim Investigational Site, A Coruña
  - 1220.30.3402 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.30.3404 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.30.3405 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.30.3408 Boehringer Ingelheim Investigational Site, Santander
  - 1220.30.3403 Boehringer Ingelheim Investigational Site, Seville
  - 1220.30.3401 Boehringer Ingelheim Investigational Site, Valencia
  - 1220.30.3407 Boehringer Ingelheim Investigational Site, Vigo (Pontevedra)
- Switzerland (5):
  - 1220.30.4106 Boehringer Ingelheim Investigational Site, Bern
  - 1220.30.4103 Boehringer Ingelheim Investigational Site, La Chaux-de-Fonds
  - 1220.30.4107 Boehringer Ingelheim Investigational Site, Lugano
  - 1220.30.4108 Boehringer Ingelheim Investigational Site, Sankt Gallen
  - 1220.30.4101 Boehringer Ingelheim Investigational Site, Zurich
- United Kingdom (9):
  - 1220.30.4405 Boehringer Ingelheim Investigational Site, Bristol
  - 1220.30.4404 Boehringer Ingelheim Investigational Site, London
  - 1220.30.4409 Boehringer Ingelheim Investigational Site, London
  - 1220.30.4410 Boehringer Ingelheim Investigational Site, London
  - 1220.30.4401 Boehringer Ingelheim Investigational Site, Manchester
  - 1220.30.4408 Boehringer Ingelheim Investigational Site, Nottingham
  - 1220.30.4407 Boehringer Ingelheim Investigational Site, Oxford
  - 1220.30.4403 Boehringer Ingelheim Investigational Site, Southampton
  - 1220.30.4406 Boehringer Ingelheim Investigational Site, Whitechapel, London

REFERENCES:
- [Derived] Jensen DM, Asselah T, Dieterich D, Foster GR, Sulkowski MS, Zeuzem S, Mantry P, Yoshida EM, Moreno C, Ouzan D, Wright M, Morano LE, Buynak R, Bourliere M, Hassanein T, Nishiguchi S, Kao JH, Omata M, Paik SW, Wong DK, Tam E, Kaita K, Feinman SV, Stern JO, Scherer J, Quinson AM, Voss F, Gallivan JP, Bocher WO, Ferenci P. Faldaprevir, pegylated interferon, and ribavirin for treatment-naive HCV genotype-1: pooled analysis of two phase 3 trials. Ann Hepatol. 2016 May-Jun;15(3):333-49. doi: 10.5604/16652681.1198803. PMID 27049487
- [Derived] Dieterich D, Nelson M, Soriano V, Arasteh K, Guardiola JM, Rockstroh JK, Bhagani S, Laguno M, Tural C, Ingiliz P, Jain MK, Stern JO, Manero M, Vinisko R, Kort J; STARTVerso4 study group. Faldaprevir and pegylated interferon alpha-2a/ribavirin in individuals co-infected with hepatitis C virus genotype-1 and HIV. AIDS. 2015 Mar 13;29(5):571-81. doi: 10.1097/QAD.0000000000000579. PMID 25710287
- [Derived] Ferenci P, Asselah T, Foster GR, Zeuzem S, Sarrazin C, Moreno C, Ouzan D, Maevskaya M, Calinas F, Morano LE, Crespo J, Dufour JF, Bourliere M, Agarwal K, Forton D, Schuchmann M, Zehnter E, Nishiguchi S, Omata M, Kukolj G, Datsenko Y, Garcia M, Scherer J, Quinson AM, Stern JO; STARTVerso1 Study Group. STARTVerso1: A randomized trial of faldaprevir plus pegylated interferon/ribavirin for chronic HCV genotype-1 infection. J Hepatol. 2015 Jun;62(6):1246-55. doi: 10.1016/j.jhep.2014.12.024. Epub 2015 Jan 2. PMID 25559324

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that they (the subject) met all strictly implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- Faldaprevir 120mg and PegIFN/RBV: Faldaprevir (BI 201335) 120 mg once daily (oral) plus Pegylated Interferon-alpha (PegIFN)/ Ribavirin (RBV) (subcutaneous injection/oral) for 12 or 24 weeks, depending on achievement of early treatment success (ETS). Patients with ETS received this treatment for 12 weeks and subsequently PegIFN/RBV alone up to Week 24; patients without ETS received this treatment for 24 weeks and subsequently PegIFN/RBV alone up to Week 48.
- Faldaprevir 240mg and PegIFN/RBV: Faldaprevir 240 mg once daily (oral) plus PegIFN/RBV (subcutaneous injection/oral) for 12 weeks, followed by PegIFN/RBV up to Week 24. Patients with ETS stopped all study medication at Week 24; patients without ETS subsequently received PegIFN/RBV alone up to Week 48.
Period: Overall Study
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Started | 259 (261 subject randomized; 259 subjects treated with at least one dose; 2 subjects were not treated) | 261 (262 subject randomized; 261 subjects treated with at least one dose; 1 subject was not treated) | 132 (133 subject randomized; 132 subjects treated with at least one dose; 1 subject was not treated)
Completed | 234 | 222 | 110
Not Completed | 25 | 39 | 22
Not completed — Adverse Event | 12 | 22 | 5
Not completed — Lack of Efficacy | 9 | 9 | 13
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 2
Not completed — other than stated above | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized patients who were dispensed study medication and were documented to have taken at least one dose.
Groups:
- Faldaprevir 120mg and PegIFN/RBV: Faldaprevir 120 mg once daily (oral) plus PegIFN/RBV (subcutaneous injection/oral) for 12 or 24 weeks, followed by PegIFN/RBV alone up to Week 24 or 48.
- Faldaprevir 240mg and PegIFN/RBV: Faldaprevir 240 mg once daily (oral) plus PegIFN/RBV (subcutaneous injection/oral) for 12 weeks, followed by PegIFN/RBV up to Week 24 or 48.
- Total: Total of all reporting groups
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV | Total
Number analyzed (Participants) | 259 | 261 | 132 | 652
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (11.44) | 48.3 (11.89) | 46.6 (12.53) | 47.8 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 115 | 57 | 310
  Male | 121 | 146 | 75 | 342

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: Sustained Virological Response 12 weeks post-treatment (SVR12), defined as plasma Hepatitis C virus (HCV) Ribonucleic acid (RNA) level < 25 IU/mL (undetected) 12 weeks after the originally planned treatment duration.
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: Full analysis set (FAS) included all randomized patients who were dispensed study medication and were documented to have taken at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
percentage of participants | 79.5 [74.6 to 84.4] | 80.5 [75.6 to 85.3] | 52.3 [43.8 to 60.8]
Statistical Analysis 1: Comparison: Faldaprevir 120mg and PegIFN/RBV vs Placebo and PegIFN/RBV; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — adjusted for genotype and race; Koch's method = 27.5, 95% CI 2-sided [17.9 to 37.0] — adjusted for genotype and race using Koch's method, with continuity correction
Statistical Analysis 2: Comparison: Faldaprevir 240mg and PegIFN/RBV vs Placebo and PegIFN/RBV; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — adjusted for genotype and race; Koch's methond = 28.6, 95% CI 2-sided [19.0 to 38.2] — adjusted for genotype and race using Koch's method, with continuity correction
Statistical Analysis 3: Comparison: Faldaprevir 120mg and PegIFN/RBV vs Faldaprevir 240mg and PegIFN/RBV; Test type: Superiority or Other; Koch's method = -1.0, 95% CI 2-sided [-7.9 to 5.8] — adjusted for genotype and race using Koch's method, with continuity correction

2. Secondary Outcome: Sustained Virological Response 24 Weeks Post-treatment (SVR24)
Description: Sustained Virological Response 24 weeks post-treatment (SVR24), defined as plasma HCV RNA level < 25 IU/mL (undetected) 24 weeks after the originally planned treatment duration.
Time Frame: 24 weeks post treatment, up to 72 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
percentage of participants | 79.2 [74.2 to 84.1] | 79.7 [74.8 to 84.6] | 52.3 [43.8 to 60.8]
Statistical Analysis 1: Comparison: Faldaprevir 120mg and PegIFN/RBV vs Placebo and PegIFN/RBV; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — adjusted for genotype and race; Koch's method = 27.1, 95% CI 2-sided [17.5 to 36.7] — adjusted for genotype and race using Koch's method, with continuity correction
Statistical Analysis 2: Comparison: Faldaprevir 240mg and PegIFN/RBV vs Placebo and PegIFN/RBV; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — adjusted for genotype and race; Koch's method = 27.8, 95% CI 2-sided [18.2 to 37.4] — adjusted for genotype and race using Koch's method, with continuity correction
Statistical Analysis 3: Comparison: Faldaprevir 120mg and PegIFN/RBV vs Faldaprevir 240mg and PegIFN/RBV; Test type: Superiority or Other; Koch's method = -0.6, 95% CI 2-sided [-7.6 to 6.3] — adjusted for genotype and race using Koch's method, with continuity correction

3. Secondary Outcome: Early Treatment Success (ETS)
Description: Early treatment success (ETS), defined as a plasma HCV RNA level <25 IU/mL (detected or undetected) at week 4 and HCV RNA <25 IU/mL (undetected) at week 8.
Time Frame: week 4 and week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
percentage of participants | 87.3 | 89.3 | 22.0

4. Secondary Outcome: Alanine Aminotransferase (ALT) Normalisation: ALT in Normal Range at End of Treatment (EoT) When SVR12=YES
Description: This will be presented as the number of patients. SVR12 means Sustained virological response 12 weeks post-treatment. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
participants
  SVR12 = Yes | 206 | 210 | 69
  SVR12 = Yes, BL normal to EoT normal | 66 | 68 | 27
  SVR12 = Yes, BL elevated to EoT normal | 97 | 115 | 31
  SVR12 = Yes, No ALT data available at EoT | 0 | 0 | 0

5. Secondary Outcome: Alanine Aminotransferase (ALT) Normalisation: ALT in Normal Range at End of Treatment (EoT) When SVR12= NO
Description: as for outcome 4
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
participants
  SVR12 = No | 53 | 51 | 63
  SVR12 = No, BL normal to EoT normal | 15 | 10 | 15
  SVR12 = No, BL elevated to EoT normal | 16 | 22 | 20
  SVR12 = No, No ALT data available at EoT | 0 | 0 | 1

6. Secondary Outcome: Alanine Aminotransferase (ALT) Normalisation: ALT in Normal Range at Sustained Virological Response 12 Weeks Post-treatment (SVR12) Visit, When SVR12=YES
Description: This will be presented as the number of patients. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
participants
  SVR12 = Yes | 206 | 210 | 69
  SVR12 = Yes, BL normal to SVR12 normal | 72 | 73 | 27
  SVR12 = Yes, BL elevated to SVR12 normal | 125 | 126 | 39
  SVR12 = Yes, No ALT data available post-treatment | 4 | 5 | 1

7. Secondary Outcome: Alanine Aminotransferase (ALT) Normalisation: ALT in Normal Range at Sustained Virological Response 12 Weeks Post-treatment (SVR12) Visit, When SVR12=NO
Description: This will be presented as the number of patients. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
participants
  SVR12 = No | 53 | 51 | 63
  SVR12 = No, BL normal to SVR12 normal | 9 | 5 | 5
  SVR12 = No, BL elevated to SVR12 normal | 6 | 6 | 1
  SVR12 = No, No ALT data available post-treatment | 8 | 14 | 45

8. Secondary Outcome: Aspartate Aminotransferase (AST) Normalisation: AST in Normal Range at End of Treatment (EoT) When SVR12=YES
Description: as for outcome 4
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
participants
  SVR12 = Yes | 206 | 210 | 69
  SVR12 = Yes, BL normal to EoT normal | 95 | 99 | 34
  SVR12 = Yes, BL elevated to EoT normal | 74 | 76 | 25
  SVR12 = Yes, No AST data available at EoT | 0 | 0 | 0

9. Secondary Outcome: Aspartate Aminotransferase (AST) Normalisation: AST in Normal Range at End of Treatment (EoT) When SVR12=NO
Description: as for outcome 4
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
participants
  SVR12 = No | 53 | 51 | 63
  SVR12 = No, BL normal to EoT normal | 17 | 16 | 21
  SVR12 = No, BL elevated to EoT normal | 14 | 16 | 13
  SVR12 = No, No AST data available at EoT | 0 | 0 | 1

10. Secondary Outcome: Aspartate Aminotransferase (AST) Normalisation: AST in Normal Range at Sustained Virological Response 12 Weeks Post-treatment (SVR12) Visit, When SVR12=YES
Description: This will be presented as the number of patients. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
participants
  SVR12 = Yes | 206 | 210 | 69
  SVR12 = Yes, BL normal to SVR12 normal | 102 | 109 | 39
  SVR12 = Yes, BL elevated to SVR12 normal | 90 | 88 | 27
  SVR12 = Yes, No AST data available post-treatment | 5 | 5 | 1

11. Secondary Outcome: Aspartate Aminotransferase (AST) Normalisation: AST in Normal Range at Sustained Virological Response 12 Weeks Post-treatment (SVR12) Visit, When SVR12=NO
Description: This will be presented as the number of patients. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 259 | 261 | 132
participants
  SVR12 = No | 53 | 51 | 63
  SVR12 = No, BL normal to SVR12 normal | 10 | 10 | 5
  SVR12 = No, BL elevated to SVR12 normal | 10 | 5 | 1
  SVR12 = No, No AST data available post-treatment | 8 | 14 | 45

ADVERSE EVENTS:
Time Frame: The double-blind treatment phase of the trial was from the randomization visit when the patient received the first dose of study drug to 30 days after the last dose of blinded trial medication up to 206 (176 +30) days.
Description: AEs that pre-existed prior to randomization but worsened during treatment were also considered treatment emergent. All patients who received at least 1 dose of study drug after randomization [safety set (SAF)] were included in the presentation of AE data.
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Serious Adverse Events (participants affected / at risk) | 17/259 | 17/261 | 8/132
Other Adverse Events (participants affected / at risk) | 246/259 | 250/261 | 120/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120mg and PegIFN/RBV (N=259) | Faldaprevir 240mg and PegIFN/RBV (N=261) | Placebo and PegIFN/RBV (N=132)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 1 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1 | 0
Retinopathy (Eye disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120mg and PegIFN/RBV (N=259) | Faldaprevir 240mg and PegIFN/RBV (N=261) | Placebo and PegIFN/RBV (N=132)
Anaemia (Blood and lymphatic system disorders) | 46 | 43 | 23
Neutropenia (Blood and lymphatic system disorders) | 32 | 25 | 18
Abdominal pain (Gastrointestinal disorders) | 11 | 15 | 10
Abdominal pain upper (Gastrointestinal disorders) | 18 | 24 | 14
Constipation (Gastrointestinal disorders) | 11 | 16 | 5
Diarrhoea (Gastrointestinal disorders) | 53 | 68 | 17
Dry mouth (Gastrointestinal disorders) | 8 | 6 | 9
Dyspepsia (Gastrointestinal disorders) | 12 | 14 | 9
Nausea (Gastrointestinal disorders) | 73 | 95 | 19
Stomatitis (Gastrointestinal disorders) | 12 | 11 | 7
Vomiting (Gastrointestinal disorders) | 28 | 52 | 6
Asthenia (General disorders) | 53 | 43 | 27
Fatigue (General disorders) | 66 | 77 | 35
Influenza like illness (General disorders) | 40 | 52 | 21
Irritability (General disorders) | 19 | 18 | 9
Malaise (General disorders) | 20 | 16 | 12
Pyrexia (General disorders) | 57 | 53 | 32
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 14 | 1
Jaundice (Hepatobiliary disorders) | 17 | 48 | 1
Nasopharyngitis (Infections and infestations) | 14 | 16 | 10
Haemoglobin decreased (Investigations) | 15 | 5 | 7
Weight decreased (Investigations) | 13 | 15 | 10
Decreased appetite (Metabolism and nutrition disorders) | 35 | 52 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 20 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 8 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 19 | 20
Disturbance in attention (Nervous system disorders) | 10 | 8 | 7
Dizziness (Nervous system disorders) | 17 | 21 | 13
Headache (Nervous system disorders) | 76 | 70 | 40
Depression (Psychiatric disorders) | 20 | 12 | 8
Insomnia (Psychiatric disorders) | 38 | 32 | 22
Sleep disorder (Psychiatric disorders) | 12 | 14 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 28 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 19 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 42 | 47 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 35 | 45 | 17
Erythema (Skin and subcutaneous tissue disorders) | 9 | 18 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 82 | 78 | 41
Rash (Skin and subcutaneous tissue disorders) | 69 | 70 | 25
Dysgeusia (Nervous system disorders) | 13 | 10 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.